CLINICAL TRIAL: NCT03159182
Title: Effectiveness of Silicone Material Inserts Within Pressure Garments in the Treatment of Hypertrophic Burn Scars
Brief Title: Study of Silicone Material Inserts To Treat Burn Scars
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: First required to complete a proof of principle study for a new outcome measure.
Sponsor: University of Manitoba (Other)
Collaborators: Health Sciences Centre Foundation, Manitoba (Other)
Responsible Party: Principal Investigator, Sara-Jane Milne, Occupational Therapist, University of Manitoba
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: B2008:056
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Burns
Keywords: Hypertrophic scarring; Silicone Material; Pressure garments
MeSH Terms: conditions — Burns; Cicatrix, Hypertrophic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pressure garment and silicone insert (Experimental): Custom measured pressure garment with a textile bonded silicone insert in either the distal or proximal portion of the pressure garment, to be worn 23 hours per day.
  Interventions: Device: Pressure garment and silicone insert
- Pressure Garment (Active Comparator): Custom measured pressure garment, to be worn 23 hours per day.
  Interventions: Device: Pressure garment

INTERVENTIONS:
Device: Pressure garment and silicone insert — Custom made fabric pressure garment with textile bonded silicone insert on either proximal or distal portion of pressure garment.
  Arms: Pressure garment and silicone insert
Device: Pressure garment — Custom made fabric pressure garment
  Arms: Pressure Garment

SUMMARY:
The purpose of this study is to determine if the use of silicone material inserts within pressure garments is effective in decreasing hypertrophic burn scar formation as compared to standard pressure garment therapy.

DETAILED DESCRIPTION:
Surgical revision, potential hospitalization, and extensive post-surgical rehabilitation may be required for the revision and correction of hypertrophic burn scars to restore function and prevent disability. This in turn results in an increased financial burden to the medical system. More importantly, the patient is required to undergo an additional invasive medical procedure that can potentially create further hypertrophic scarring.

Prevention and reduction of hypertrophic scars with non-invasive, cost effective, and evidence based treatment modalities is therefore the most desirable approach. Two of the most generally accepted methods of non-invasive treatment, pressure garments and silicone gel sheeting, have been demonstrated to individually treat hypertrophic scarring. Recently, burn therapists have begun to use silicone bonded material inserts within pressure garments following the logical deduction that the two therapeutic techniques can be combined to resolve many of the cited individual disadvantages, while reaping the benefits of each individual modality. It is the aim of this study to determine the efficacy of these silicone bonded material inserts within pressure garments in the treatment of hypertrophic scarring.

ELIGIBILITY:
Inclusion Criteria:

* patients who would normally receive pressure garments
* presence of an acute burn to an upper or lower extremity that requires treatment with a sheet or meshed graft
* Minimum 4% total body surface area graft dimension (this must include areas above and below the elbow or on medial and lateral aspects of the calf
* Between 16 years and 60 years of age
* Patient must consent to the study or obtain consent from guardian if <18 years of age
* Must be available for follow-up at 1 month, 3 months, 6 months, and 12 months post initiation of treatment

Exclusion Criteria:

* Presence of pre-existing hypertrophic or keloid scarring
* Pressure garments initiated greater than 2 months post discharge from hospital
* Pre-existing decrease in range of motion of affected extremity
* One treatment area with a prolonged healing phase or which had been treated differently in comparison to adjacent treatment area
* Patient unable to comprehend or participate in self reporting

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Scar pliability measured in gm/mm squared | A baseline evaluation will be performed at the time of initial pressure garment fitting, and follow up evaluations will take place at 1 month, 3 months, 6 months and 12 months after pressure garment fitting.
  The Modified Vancouver Scar Scale (MVSS) will be used to measure the scar pliability. It is a therapist-judged hand held tool that measure scar properties on an ordinal scale. Because the MVSS is a subjective rating system, we will also be using the NK Skin Compliance Device (SCD)to measure scar pliability. It is a non-invasive hand-held device that measures skin compliance or pliability.

SECONDARY OUTCOMES:
Scar vascularity | A baseline evaluation will be performed at the time of initial pressure garment fitting, and follow up evaluations will take place at 1 month, 3 months, 6 months and 12 months after pressure garment fitting.
  The Modified Vancouver Scar Scale (MVSS) will be used to measure the scar pliability. It is a therapist-judged hand held tool that measure scar properties on an ordinal scale.

OTHER OUTCOMES:
Scar height | A baseline evaluation will be performed at the time of initial pressure garment fitting, and follow up evaluations will take place at 1 month, 3 months, 6 months and 12 months after pressure garment fitting.
  The Modified Vancouver Scar Scale (MVSS) will be used to measure the scar pliability. It is a therapist-judged hand held tool that measure scar properties on an ordinal scale.
Scar itch | A baseline evaluation will be performed at the time of initial pressure garment fitting, and follow up evaluations will take place at 1 month, 3 months, 6 months and 12 months after pressure garment fitting.
  Scar itch will be measured using a visual analogue scale (VAS).
Scar Appearance | A baseline evaluation will be performed at the time of initial pressure garment fitting, and follow up evaluations will take place at 1 month, 3 months, 6 months and 12 months after pressure garment fitting.
  Will be measured using a visual analogue scale (VAS).
Comfort of garment | A baseline evaluation will be performed at the time of initial pressure garment fitting, and follow up evaluations will take place at 1 month, 3 months, 6 months and 12 months after pressure garment fitting.
  Will be measured using ordered response scales.
Limitations to movement | A baseline evaluation will be performed at the time of initial pressure garment fitting, and follow up evaluations will take place at 1 month, 3 months, 6 months and 12 months after pressure garment fitting.
  Will be measured using ordered response scales.

CONTACTS AND LOCATIONS:
Overall Officials: Sara-Jane Milne, BMR(OT), Principal Investigator — Winnipeg Health Sciences Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baryza MJ, Baryza GA. The Vancouver Scar Scale: an administration tool and its interrater reliability. J Burn Care Rehabil. 1995 Sep-Oct;16(5):535-8. doi: 10.1097/00004630-199509000-00013. PMID 8537427
- [Result] Ahn ST, Monafo WW, Mustoe TA. Topical silicone gel: a new treatment for hypertrophic scars. Surgery. 1989 Oct;106(4):781-6; discussion 786-7. PMID 2529659
- [Result] Allely RR, Van-Buendia LB, Jeng JC, White P, Wu J, Niszczak J, Jordan MH. Laser Doppler imaging of cutaneous blood flow through transparent face masks: a necessary preamble to computer-controlled rapid prototyping fabrication with submillimeter precision. J Burn Care Res. 2008 Jan-Feb;29(1):42-8. doi: 10.1097/BCR.0b013e31815f6eeb. PMID 18182896
- [Result] Al-Mandeel, MS, Bang, R.L., & Ebrahim, M.K. Re-appraisal of cica-care (silicone gel sheet) in ther treatment of hypertrophic and keloid scars. Saudi Medical Journal 19(6):741-745, 1998.
- [Result] Bartell TH, Monafo WW, Mustoe TA. A new instrument for serial measurements of elasticity in hypertrophic scar. J Burn Care Rehabil. 1988 Nov-Dec;9(6):657-60. doi: 10.1097/00004630-198811000-00021. PMID 3220875
- [Result] Baur PS, Larson DL, Stacey TR, Barratt GF, Dobrkovsky M. Ultrastructural analysis of pressure-treated human hypertrophic scars. J Trauma. 1976 Dec;16(12):958-67. doi: 10.1097/00005373-197612000-00004. No abstract available. PMID 1003586